CLINICAL TRIAL: NCT00643968
Title: Randomized Multicenter Open-Label, Pilot Trial to Evaluate the Efficacy and Safety of Switching HIV-1 Stable Infected Patients Under HAART to a New Once Daily Triple Therapy Combination Including EFV+3TC+TDF Versus a Dual QD Therapy Containing EFV+TDF
Brief Title: Tenofovir DF + Efavirenz (TDF+EFV) Versus Tenofovir DF + Efavirenz + Lamivudine (TDF+EFV+3TC) Maintenance Regimen in Virologically Controlled Patients: COOL Trial
Acronym: COOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Dr Aldo Trylesinski- Gilead Sciences, Gilead Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GS-FR-104-1016
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV virological control; Lipid profile and morphological fat distribution; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): TDF+EFV
  Interventions: Drug: EFV+TDF
- 2 (Experimental): TDF+3TC+EFV
  Interventions: Drug: EFV+3TC+TDF

INTERVENTIONS:
Drug: EFV+TDF
  Arms: 1
Drug: EFV+3TC+TDF
  Arms: 2

SUMMARY:
Primary objective: Evaluation of the efficacy of TDF+3TC+EFV versus TDF+EFV QD to maintain plasma HIV-1 RNA BLQ (< 50 copies/mL) (c/mL) at 48 weeks (W48)

Main Secondary objectives:

Comparison of the two arms for genotypic resistance profile in case of virological failure

CD4 changes from baseline

Evolution of the lipid profile and morphological changes in fat distribution, and safety

Efficacy and genotypic profile data, results of lipid markers, morphological changes and main biological parameters

ELIGIBILITY:
Inclusion Criteria:

* Stable HAART ≥ 3 months
* HIV-1 RNA < 50 c/mL ≥ 6 months
* No HAART failure history

Exclusion Criteria:

* Weight > 45 kg
* No CD4+ cell count criteria
* No significant laboratory or clinical abnormalities
* Creatinine Clearance > 60 mL/min

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-03; Primary Completion 2005-06 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of TDF+3TC+EFV versus TDF+EFV QD to maintain plasma HIV-1 RNA BLQ (< 50 copies/mL) (c/mL) at 48 weeks (W48) | 48 wks

SECONDARY OUTCOMES:
Comparison of the two arms for genotypic resistance profile in case of virological failure | 48 wks
CD4 changes from baseline | 48 wks
Evolution of the lipid profile and morphological changes in fat distribution, and safety | 48 wks

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Trylesinski, MD, Principal Investigator — Gilead Sciences
Locations (1):
- France and French West Indies, Paris, France

REFERENCES:
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-02-1016_synopsis.pdf